CLINICAL TRIAL: NCT00178958
Title: Evaluation of QTc Interval by Continuous Holter ECG Recording in Antipsychotic Drug-treated Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Herbert Meltzer, Professor, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 030459
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Schizoaffective; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Holter Monitor

SUMMARY:
The aim of this study is to evaluate the utility of continuous Holter ECG recording with automated, computerized data analysis for measuring antipsychotic-related QTc prolongation during a 24-h period under clinical conditions

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males or females between 18 - 65 years of age.
2. Patient subjects will have a definite diagnosis by DSM-IV criteria, schizophrenia, schizoaffective disorder, or bipolar disorder.
3. Patient subjects are currently under treatment with any antipsychotic, any mood stabilizer, any antidepressant or any combination of the above at the therapeutic dose for at least 3 months.
4. Patients have a history of taking the medications listed in item 3 as prescribed.
5. The subjects must be able to provide written informed consent

Exclusion Criteria:

1. Subjects with a DSM-IV diagnosis of substance dependence as defined by DSMN within three months prior to selection.
2. Subjects who are currently taking other medications that have been shown to prolong the QTc, including tricyclic antidepressants (e.g. amitriptyline, imipramine, maprotiline), fluoroquinolones, or antiarrhythmics (e.g. quinidine, procainamide, amiodarone, sotalol).

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to evaluate the utility of continuous Holter ECG recording with automated, computerized data analysis for measuring antipsychotic-related QTc prolongation during a 24-h period under clinical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center